CLINICAL TRIAL: NCT05090735
Title: Are Superficial Parasternal Intercostal Plane (SPIP) Blocks With Transversus Abdominis Plane (TAP) Block More Helpful Than SPIP Blocks Alone in Managing Post-operative Pain in Coronary Artery Bypass Grafting (CABG)?
Brief Title: Are Superficial Parasternal Intercostal Plane (SPIP) Blocks With Bupivacaine and With or Without Transversus Abdominis Plane Block (TAP) Helpful for Post-operative Pain After Coronary Artery Bypass Grafting?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Sandeep Krishnan, Associate Professor of Anesthesiology, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SPIP and TAP in CABG
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Post-operative Pain Management
Keywords: coronary artery bypass grafting, superficial parasternal intercostal plane block , transversus abdominis plane block, opioid consumption

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPIP Block (Active Comparator): 50 Patients-Post-operatively patients will receive bilateral SPIP blocks by injecting 20 mL of 0.25% bupivacaine (on each side) between the pectoralis major and external intercostal muscle aponeurosis at 2 cm lateral to the right and left of the sternal edge, corresponding to the fifth rib.
  Interventions: Procedure: SPIP Block
- SPIP Block with TAP Block (Active Comparator): 50 Patients-Post-operatively patients will receive bilateral SPIP blocks by injecting 20 mL of 0.25% bupivacaine (on each side) between the pectoralis major and external intercostal muscle aponeurosis at 2 cm lateral to the right and left of the sternal edge, corresponding to the fifth rib. This group of patients will also receive unilateral TAP block by injecting 20 mL of 0.25% bupivacaine in the plane between the internal oblique and transversus abdominis muscles.
  Interventions: Procedure: SPIP and TAP Block

INTERVENTIONS:
Procedure: SPIP and TAP Block — Injection of Bupivacaine 0.25% for SPIP Block and TAP Block.
  Arms: SPIP Block with TAP Block
Procedure: SPIP Block — Injection of Bupivacaine 0.25% for SPIP Block
  Arms: SPIP Block

SUMMARY:
The purpose of this study is to determine whether superficial parasternal intercostal plane (SPIP) block alone or with transverses abdominis plane (TAP) block can improve post-operative pain in patients undergoing cardiothoracic surgery, specifically, coronary artery bypass grafting (CABG).

DETAILED DESCRIPTION:
Postoperative pain management remains an important clinical challenge in cardiothoracic surgery. Inadequate postoperative pain control can have adverse pathophysiologic consequences, including increased myocardial oxygen demand, hypoventilation, suboptimal clearance of pulmonary secretions, acute respiratory failure, and decreased mobility, with associated increased risks for formation of clots in a blood vessels (thromboembolism). These adverse events may result in greater perioperative morbidity and mortality. Despite several multimodal approaches to postoperative pain control, optimal pain management after cardiothoracic procedures remains an issue.

Regional anesthesia is used to block sensation in a specific part of body during and after surgery. It offers numerous advantages over conventional general anesthesia, including faster recovery time, fewer side effects, no need for an airway device during surgery, and a dramatic reduction in post-surgical pain and reduction in opioid use following surgery. The use of local anesthetic peripheral nerve blocks for surgical anesthesia and postoperative pain management has increased significantly with the advent of ultrasound-guided techniques.

Ultrasound has revolutionized regional anesthesia by allowing real-time visualization of anatomical structures, needle advancement and local anesthetic (LA) spread. This has led not only to refinement of existing techniques, but also the introduction of new ones.

In particular, ultrasound has been critical in the development of fascial plane blocks, in which local anesthetic (LA) is injected into a tissue plane rather than directly around nerves. These blocks are believed to work via passive spread of LA to nerves traveling within that tissue plane, or to adjacent tissue compartments containing nerves.

Although research into these techniques is still at an early stage, the available evidence indicates that they are effective in reducing opioid requirements and improving the pain experience in a wide range of clinical settings. They are best employed as part of multimodal analgesia with other systemic analgesics, rather than as sole anesthetic techniques. Catheters may be beneficial in situations where moderate-severe pain is expected for >12 hours, although the optimal dosing regimen requires further investigation.

In this study the investigators will focus on the superficial parasternal-intercostal plane (SPIP) block and the transverses abdomens plane (TAP) block.

The investigators will compare the SPIP block administered alone and with a TAP block; the investigators will measure the visual analog scale (VAS) pain scores in the first 24 hours after surgery, total post-operative opioid consumption (oral morphine equivalents), total acetaminophen and ketorolac consumption, post-operative nausea and vomiting (PONV), length of the ICU stay, time to extubation, and length of hospital stay to determine if one technique is superior to the other.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing primary coronary artery bypass grafting

Exclusion Criteria:

* Patients with significant genetic or acquired clotting/bleeding disorders (hemophilia, DIC, etc.)
* Patients with significant platelet dysfunction
* Infection at site for regional anesthesia
* Allergy to local anesthetics
* Severe aortic stenosis
* Severe mitral stenosis
* Sepsis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Post-operative total opioid consumption (oral morphine equivalents) | 24 hours after surgery
  Total Opioid consumption 24 hours post surgery oral moral morphine equivalents
Visual analog scale (VAS) pain scores | 6 hours after surgery
  Pain Scores measured via a Visual Analog Scale (0-10, Higher scores mean worse outcome)
Visual analog scale (VAS) pain scores | 12 hours after surgery
  Pain Scores measured via a Visual Analog Scale (0-10, Higher scores mean worse outcome)
Visual analog scale (VAS) pain scores | 24 hours after surgery
  Pain Scores measured via a Visual Analog Scale (0-10, Higher scores mean worse outcome)
Length of hospital stay (LOS) | Up to 1 month
  The days spent in the hospital from surgery to discharge

SECONDARY OUTCOMES:
Incidence of post-operation nausea and vomiting (PONV) | 24 hours
  The percentage of the patients who had post-operative nausea and vomiting (PONV) within 24 hours of surgery
Acetaminophen consumption | 24 hours after surgery
  Total acetaminophen consumption in mg 24 hr after surgery
NSAID (ketorolac) consumption | 24 hours after surgery
  Total NSAID consumption in mg
Length of ICU stay | Up to 1 month
  Length of stay in Intensive Care Unit from surgery to discharge from Intensive Care Unit
Time to extubation | 24 hours
  Time it took for patient to be extubated

IPD SHARING:
Plan to Share IPD: No